CLINICAL TRIAL: NCT06680024
Title: Comparative Study Between Outcome of Inter-costal Tube Drainage and Video Assisted Thoracoscopic Surgery in Management of Second Stage Empyema
Brief Title: Comparative Study Between Outcome of ICT Drainage and VATS in Management of Second Stage Empyema
Acronym: ICT and VATS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Sayed Khalaf, Resident at cardiothoracic surgery department, sohag university hospitals, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-24-09-10MS
Record Dates: First submitted 2024-11-05; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-09

CONDITIONS: Second Stage Empyema
MeSH Terms: interventions — Chest Tubes; Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intercostal tube (Active Comparator): Intercostal tube as a primary intervention for treatment of second stage empyema
  Interventions: Procedure: Intercostal tube
- Video assisted thoracoscope (Active Comparator): Video assisted thoracoscopic evacuation as a primary intervention for treatment of nd stage empyema
  Interventions: Procedure: Video assisted thoracoscope

INTERVENTIONS:
Procedure: Intercostal tube — Intercostal tube drainage as a first management of second stage empyema
  Other Names: Chest tube
  Arms: Intercostal tube
Procedure: Video assisted thoracoscope — Video assisted thoracoscopic surgery as a first management for second stage empyema
  Other Names: VATS
  Arms: Video assisted thoracoscope

SUMMARY:
The goal of this clinical trial is to compare between outcome of inter-costal tube drainage and video assisted thoracoscopic surgery in management of patients with second stage empyema.

It compares the outcome of both interventions in hospital stay, cost, wether need of decortication later on or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients both adults and children diagnosed as Empyema thoracis in early stages based on clinical examination, imaging modalities and pleural fluid analysis

Exclusion Criteria:

* Empyema due to carcinoma, terminally ill patients, patients with severe respiratory distress at admission, patients not fit for surgery, patients with co morbid diseases like cardiac disorders and immunosuppression.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-10 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
the length of hospital stay | From enrollment to 4 weeks
  Comparison between both intercostal tube drainage and video assisted thoracoscopic surgery in management of patients with second stage empyema, we will compare the length of hospital stay of each group of patients
cost of treatment of the patients' in each group | 4 weeks
  Comparison between both intercostal tube drainage and video assisted thoracoscopic surgery in management of patients with second stage empyema, we will compare cost of treatment of the patients' in each group
number of participants with needs of decortication later on or not, assessed by the chest X-ray and CT chest. | 4 weeks
  Comparison between both intercostal tube drainage and video assisted thoracoscopic surgery in management of patients with second stage empyema, we will compare with the chest X-ray and CT chest if there is residual empyema and whether the patients will need decortication later on or not

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/18570573/
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC3919299/